CLINICAL TRIAL: NCT00259961
Title: Clinical Outcome of Laparoscopic Versus Open Nissen Fundoplication in Children: 3-Year Follow-up Study of Randomized Controlled Trial.
Status: Completed | Type: Observational
Sponsor: Institute of Child Health (Other)
Other Study IDs: 05SG29
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Gastro -Oesophagal Reflux

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: open fundoplication
Procedure: laparoscopic fundopliaction

SUMMARY:
Long-term results following laparoscopic and open Nissen fundoplication for gastro-oesophageal reflux will be objectively assessed in a selected population of patients already included in a randomized controlled trial comparing the two different techniques. The presence of postoperative symptoms will be evaluated by an independent clinician using an objective questionnaire. The recurrence of gastro-oesophageal reflux will be studied by 24-hours pH study. Furthermore the presence of gastric motility disorders will be studied by electrogastrography and 13C-octanoic acid breath test.

ELIGIBILITY:
Inclusion Criteria: All patients with gastro - oesophagal reflux -

Exclusion Criteria:

-

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Pierro Agostino, Prof, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Pacilli M, Eaton S, McHoney M, Kiely EM, Drake DP, Curry JI, Lindley KJ, Pierro A. Four year follow-up of a randomised controlled trial comparing open and laparoscopic Nissen fundoplication in children. Arch Dis Child. 2014 Jun;99(6):516-21. doi: 10.1136/archdischild-2013-304279. Epub 2014 Feb 14. PMID 24532685